CLINICAL TRIAL: NCT06188182
Title: D-index as a Predictor of Complications of Febrile Neutropenia in Patients With Acute Myeloid Leukemia
Brief Title: D-index as a Predictor of Complication of Treatment of Patients With Acute Myeloid Leukemia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Nageh Adam, Assistant Lecture, Assiut University
Other Study IDs: neutropnic fever in AML
Record Dates: First submitted 2023-12-14; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. The effect of D-index on the onset and severity of FN in AML patients.
2. Relationship between the c-D-index and duration of FN in AML patients.
3. Correlation between D-index and MDR.
4. Correlation between D-index and invasive fungal infection.
5. Comparison of FN in different treatment protocols for AML using D-index.
6. Prediction of pulmonary, fungal or blood stream infection.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is highly malignant neoplasm responsible for a large number of cancer-related deaths. It continuously shows 2 peaks in occurrence in early childhood and later adulthood. With an incidence of 3.7 per 100,000 persons per year.

Neutropenia, defined as the absolute neutrophil count (ANC) below 500 cells/ μL or ANC expected to drop below 500 cells/ μL in the next 48 h, represents a potentially fatal complication and is associated with a high risk of developing bacterial infections. Fever is defined as having a bodily temperature above 38.3 ˚C, measured orally, or two measurements above 38 ˚C that are taken at different time points, at least an hour apart.

Concomitance of severe neutropenia (≤ 500 cells/ μL) with high fever (≥ 38.3˚C) is called febrile neutropenia (FN) by the definition of the Infectious Diseases Society of America (IDSA).

Invasive fungal infection (IFI) and bacterial blood stream infection (BSI) consideded a major complications during AML treatment and associated with high morbidity and mortality. Immunosuppression caused by chemotherapy and prolonged hospitalizations expose AML patients to life threatening infections, which can be sustained by multi-drug resistant organisms (MDROs), accounting for one of the major causes of mortality.

A clinical parameter that evaluates the dynamics of neutropenia, combining intensity and duration, could be a good tool to identify patients at high risk for infection. This tool could be used to stratify patients, helping clinicians to select appropriate antibiotics and antifungal therapy in persistently febrile neutropenic patients. An index (called the D-index) that uses data from WBC counts and combines intensity and duration of neutropenia.

The D-index was developed by the calculated area over the neutrophil curve from the plot of ANC<500 /μl and duration of grade 4 neutropenia. Cumulative D-index (c-D-index) was also defined from the grade 4 neutropenia to the onset of febrile neutropenia, it reflects an accumulation of neutropenia until FN. Therefore, this study aim to describe and investigate the impacts of D-index performance on infectious complications in adult AML patients who developed the first episode of FN after receiving high-intensity chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients (≥18 years) newly diagnosed as acute myeloid leukemia according to WHO 2016 diagnostic criteria.
2. Hematologic diagnosis of de novo AML.
3. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2.
4. Standard induction chemotherapy (7+3 regimen) or consolidation regimens (HiDAC).

Exclusion Criteria:

1) AML on top of other hematological disorders. 2) Acute promyelocytic leukemia. 3) Patients who received palliative care or low-intensity treatment. 4) Poor PS (≥3) at the time of diagnosis.

-

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients meeting the inclusion criteria will be recruited in the study. The period of data collection will be continued for 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The effect of D-index on the onset and severity of FN in AML patients. | during the period of chemotherapy completion, an average of 1 year
  Determine if the D-index can predict the onset, severity, duration and complications of febrile neutropenia

REFERENCES:
- [Result] Deschler B, Lubbert M. Acute myeloid leukemia: epidemiology and etiology. Cancer. 2006 Nov 1;107(9):2099-107. doi: 10.1002/cncr.22233. PMID 17019734
- [Result] Boeriu E, Borda A, Vulcanescu DD, Sarbu V, Arghirescu ST, Ciorica O, Bratosin F, Marincu I, Horhat FG. Diagnosis and Management of Febrile Neutropenia in Pediatric Oncology Patients-A Systematic Review. Diagnostics (Basel). 2022 Jul 25;12(8):1800. doi: 10.3390/diagnostics12081800. PMID 35892511
- [Result] Freifeld AG, Bow EJ, Sepkowitz KA, Boeckh MJ, Ito JI, Mullen CA, Raad II, Rolston KV, Young JA, Wingard JR; Infectious Diseases Society of Americaa. Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2011 Feb 15;52(4):427-31. doi: 10.1093/cid/ciq147. Epub 2011 Jan 4. PMID 21205990
- [Result] Amanati A, Sajedianfard S, Khajeh S, Ghasempour S, Mehrangiz S, Nematolahi S, Shahhosein Z. Bloodstream infections in adult patients with malignancy, epidemiology, microbiology, and risk factors associated with mortality and multi-drug resistance. BMC Infect Dis. 2021 Jul 2;21(1):636. doi: 10.1186/s12879-021-06243-z. PMID 34215207
- [Result] Guarnera L, Trotta GE, Boldrini V, Cardillo L, Cerroni I, Mezzanotte V, Pasqualone G, Savi A, Borsellino B, Buzzatti E, Palmieri R, Paterno G, Maurillo L, Buccisano F, Venditti A, Del Principe MI. Fever of Unknown Origin and Multidrug Resistant Organism Colonization in AML Patients. Mediterr J Hematol Infect Dis. 2023 Jan 1;15(1):e2023013. doi: 10.4084/MJHID.2023.013. eCollection 2023. PMID 36660358
- [Result] Rattanathammethee T, Munsamai K, Punnachet T, Hantrakun N, Piriyakhuntorn P, Hantrakool S, Chai-Adisaksopha C, Rattarittamrong E, Tantiworawit A, Norasetthada L. D-index and invasive fungal infections (IFIs) in adult acute myeloid leukemia (AML) patients with the first episode of febrile neutropenia. PLoS One. 2023 May 22;18(5):e0286089. doi: 10.1371/journal.pone.0286089. eCollection 2023. PMID 37216345
- [Result] Portugal RD, Garnica M, Nucci M. Index to predict invasive mold infection in high-risk neutropenic patients based on the area over the neutrophil curve. J Clin Oncol. 2009 Aug 10;27(23):3849-54. doi: 10.1200/JCO.2008.21.0856. Epub 2009 Jul 13. PMID 19597026